CLINICAL TRIAL: NCT06838078
Title: Evaluation of the Trend Correlation Between End-Tidal and Arterial Carbon Dioxide Partial Pressures During Laparoscopic Surgery in the Trendelenburg Position: A Prospective Observational Study
Brief Title: Trend Correlation Between End-Tidal and Arterial Carbon Dioxide During Laparoscopic Surgery in Trendelenburg Position
Status: Not yet recruiting | Type: Observational
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Kamil Darcin, Associate Professor, Koç University
Other Study IDs: 2024.271.IRB1.035
Record Dates: First submitted 2025-02-12; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Laparoscopic Surgery; Trendelenburg Position

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, we want to find out whether a person's "end-tidal carbon dioxide" (ETCO₂)-a value measured from the air they breathe out-accurately reflects the amount of carbon dioxide in their blood, called "arterial carbon dioxide" (PaCO₂).

We are focusing on people having laparoscopic (keyhole) surgery in the Trendelenburg position, which involves tilting the patient's head down to help the surgeon see the surgical area better. This position can sometimes affect carbon dioxide levels in the blood. Right now, doctors must draw blood samples to measure the PaCO₂ level. If we can show that ETCO₂ readings are reliable, doctors may not need to draw blood samples as often.

During surgery, patients already need a small tube (catheter) in an artery so doctors can closely monitor their blood pressure. Whenever the anesthesiologist decides a blood sample is needed, we will note the blood's PaCO₂ level and compare it with the ETCO₂ reading taken at the same time. We will also record other measurements like heart rate, blood pressure, and temperature.

By comparing these measurements, we hope to learn if the ETCO₂ readings can reliably match the changes in PaCO₂ over time, making it a useful tool to monitor carbon dioxide levels in this type of surgery without needing as many blood tests. We plan to include 79 patients in this study, which should give us enough measurements to see how closely these two methods match.

DETAILED DESCRIPTION:
Laparoscopic surgeries performed in the Trendelenburg position require tilting the patient's head downward, which can help provide optimal visualization of the surgical field. However, this position may increase intrathoracic pressure and reduce venous return, leading to potential changes in arterial carbon dioxide (PaCO₂) levels. Arterial blood gas (ABG) sampling remains the gold standard for measuring PaCO₂, but it is invasive, costly, and provides only intermittent data. End-tidal carbon dioxide (ETCO₂) monitoring, available through standard anesthesia devices, offers continuous, noninvasive measurement of exhaled CO₂ and can serve as a surrogate for PaCO₂.

The primary purpose of this study is to evaluate the agreement and trend correlation between ETCO₂ and PaCO₂ in patients undergoing laparoscopic procedures in the Trendelenburg position. If ETCO₂ reliably tracks changes in PaCO₂, clinicians may safely reduce the number of ABG samples required during these operations, minimizing patient discomfort and healthcare costs.

Primary objective: To evaluate the trend correlation between ETCO₂ and PaCO₂ over time using four-quadrant and polar plot analyses.

Secondary objective: To determine the degree of agreement between ETCO₂ and PaCO₂

Study Type: Prospective, observational study. Study Setting: Operating rooms where adult patients (≥18 years old) are scheduled for laparoscopic surgery in the Trendelenburg position and require invasive arterial pressure monitoring as part of their routine care.

Duration: Each patient's participation will be limited to the intraoperative period (i.e., from anesthesia induction to the end of surgery).

Intraoperative management will follow a standardized anesthetic protocol, and ABG samples will be drawn at the anesthesiologist's discretion whenever clinically indicated.

Each time an ABG is taken, the corresponding ETCO₂, PaCO₂, arterial blood pressure, heart rate, and temperature values will be recorded.

Any use of inotropic or antihypertensive infusions will be documented, as such medications can influence hemodynamic stability and possibly ventilatory parameters.

The patient's demographic details (age, sex, height, weight) and the type of surgical procedure will be recorded.

Four-quadrant and polar plots will be generated to assess the concordance of changes in ETCO₂ with changes in PaCO₂ over time.

Bland-Altman plots will be constructed to calculate the mean difference (bias) and 95% limits of agreement for each paired measurement.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo laparoscopic surgery in the Trendelenburg position
* Planned to receive invasive arterial blood pressure monitoring as part of routine clinical care (independent of the study)

Exclusion Criteria:

* Chronic obstructive pulmonary disease
* Pulmonary hypertension
* Active systemic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be drawn from the adult patient population (≥18 years) scheduled for laparoscopic surgery in the Trendelenburg position at a tertiary care hospital. These individuals are already indicated to receive invasive arterial blood pressure monitoring as part of their routine clinical management. No special outreach or community recruitment methods will be employed; rather, eligible patients will be identified from the hospital's surgical wards and preoperative clinics.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Trend correlation between ETCO₂ and PaCO₂ measured by the concordance ratio in the four-quadrant plot | During the surgery of the patient, arterial blood gas samples will be drawn at the anesthesiologist's discretion whenever clinically indicated.
  A four-quadrant plot will be generated by comparing consecutive changes (deltas) in PaCO₂ and ETCO₂. For each patient, every pair of sequential measurements will be used to calculate ΔPaCO₂ (horizontal axis) and ΔETCO₂ (vertical axis). Points in the top-right (Quadrant I) and bottom-left (Quadrant III) indicate concordant changes (both variables increased or both decreased). A "central zone" will be defined to exclude clinically negligible fluctuations (±1mmHg). The percentage of points in Quadrant I and III, relative to those outside the central zone, will be reported as the overall concordance. A concordance ratio above 90% will be considered as good trending ability.
Trend correlation between ETCO₂ and PaCO₂ measured by the angular bias in the four-quadrant plot | During the surgery of the patient, arterial blood gas samples will be drawn at the anesthesiologist's discretion whenever clinically indicated.
  In the four-quadrant plot, the angle of each data point relative to the 45-degree line will be calculated. The average of this angles will be reported as angular bias. An angular bias between ±5 degrees will be considered as good trending ability.
Trend correlation between ETCO₂ and PaCO₂ measured by radial limits of aggreement in the four-quadrant plot | During the surgery of the patient, arterial blood gas samples will be drawn at the anesthesiologist's discretion whenever clinically indicated.
  In the four-quadrant plot, the angle of each data point relative to the 45-degree line will be calculated. The radial sector that contains 95% of the data points will be reported as radial limits of agreement. Radial limits of agreement between ±30 degrees will be considered as good trending ability.

SECONDARY OUTCOMES:
Aggreement between simultaneous ETCO₂ and PaCO₂ values measured by limits of aggreement in Bland-Altman plot | During the surgery of the patient, arterial blood gas samples will be drawn at the anesthesiologist's discretion whenever clinically indicated.
  A Bland-Altman plot will be used to assess agreement between ETCO₂ and PaCO₂. For each paired measurement, the difference between ETCO₂ and PaCO₂, and the average of ETCO₂ and PaCO₂ will be calculated. Each point will be plotted with the difference on the vertical axis against the average on the horizontal axis. The mean difference (bias) and 95% limits of agreement (mean difference ± 1.96 × SD of the difference) will then be calculated. Limits of aggreement between ±4 mmHg will be considered as good aggreement.